CLINICAL TRIAL: NCT06717412
Title: Efficacy and Safety of Low-dose Conbercept for Retinopathy of Prematurity Therapy: A Multicenter, Prospective, Randomized, Double-blind, Non-inferiority Clinical Trial
Brief Title: Efficacy and Safety of Low-dose Conbercept for Retinopathy of Prematurity Therapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wang Yusheng (Other)
Responsible Party: Sponsor-Investigator, Wang Yusheng, Professor, Xijing Hospital
Organization: Xijing Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KY20242291
Record Dates: First submitted 2024-11-28; First posted 2024-12-05 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2024-11

CONDITIONS: Retinopathy of Prematurity (ROP)
MeSH Terms: conditions — Retinopathy of Prematurity | interventions — KH902 fusion protein

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Conbercept 0.25 mg/0.025mL (Active Comparator): intravitreal injection in both eyes on Day 0, with up to 1 re-treatment allowed for each eye if required
  Interventions: Drug: Conbercept
- Conbercept 0.15 mg/0.015mL (Experimental): intravitreal injection in both eyes on Day 0, with up to 1 re-treatment allowed for each eye if required
  Interventions: Drug: Conbercept

INTERVENTIONS:
Drug: Conbercept — Administered as an intravitreal injection

SUMMARY:
Evaluating the Optimal Effective Dose and Safety of Conbercept in Treating Retinopathy of Prematurity (ROP)

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants with less than or equal to 2000 grams of birth weight or less than or equal to 32 weeks of gestational age
* Bilateral type 1 ROP with one of the following retinal findings in each eye
* Zone I, stage 1+, 2+, 3+/- disease, or
* Zone II, stage 2+, 3+, disease, or
* A-ROP

Exclusion Criteria:

* Preterm infants with stage 4 or 5 ROP in one or both eyes
* Have received any previous surgical or nonsurgical treatment for ROP, including laser photocoagulation, anti-VEGF therapy, vitrectomy
* Have been previously exposed to any intravitreal or systemic anti-VEGF agent (either the patient or the mother during this child's pregnancy)
* Have used (either the patient or the mother) other investigational drugs as part of another clinical study (other than vitamins and minerals) within 30 days or within 5 half-lives of the other investigational drug, whichever is longer
* Have active ocular infection within 5 days before or on the day of first investigational treatment
* Have a history of hypersensitivity (either the patient or the mother) to any of the investigational treatments or to drugs of similar chemical classes
* Have any contraindication for intravitreal injection clearly stated in the instructions
* Have any ocular structural abnormality that may affect efficacy assessments
* Have a history of any other congenital or systemic conditions that are assessed by the investigator to have a significant risk of severe impact on visual function
* Have any other medical conditions or clinically significant comorbidities or personal circumstances that are assessed by the investigator to have a clinically relevant impact on study participation, any of the study procedures, or on efficacy assessments

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 146 (Estimated)
Dates: Start 2024-11-29 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with absence of active ROP and absence of unfavorable structural outcomes in both eyes during the observational period after starting study treatment | Week 24
  To achieve this outcome, participants cannot fulfill any of the following criteria:
  1. Require intervention for ROP in either eye at or before the week 24 assessment visit with a treatment modality other than Conbercept
  2. Have active ROP in either eye at the week 24 assessment visit
  3. Have unfavorable structural outcomes (e.g., retinal detachment, retinal traction, macular abnormalities) in either eye at or before week 24 assessment visit

SECONDARY OUTCOMES:
Percentage of participants with effective single intravitreal injection treatment | Week 24
  Effective single intravitreal injection treatment is defined as regression of ridge and plus disease after the first study treatment.
Percentage of participants having reactivation at or before week 24 | Week 24
  Reactivation of ROP is defined as ridge-like change or fibrovascular proliferation occur at the original lesion site, accompanied by the reappearance of plus disease.
Percentage of participants with complete vascularization of the peripheral retina at or before week 24 | Week 24
  Complete vascularization is defined as participants fulfill any of the following criteria:
  1. Fundus photography shows the temporal vessels are less than 2 disc diameter from the ora serrata or the nasal vessels are less than 1 disc diameter from the ora serrata
  2. Fluorescein fundus angiography shows the ratio of the distance from the center of the disk to the border of the vascularized zone (DB) and the distance from the center of the disk to the center of the fovea (DF) is greater than 4.0 temporally or greater than 3.3 nasally
Percentage of participants requiring repeated intervention at or before week 24 | Week 24
  Repeated intervention is defined as receiving other intervention after the first treatment, regardless of the modality.
Percentage of participants requiring interventions with a second modality for ROP at or before week 24 | Week 24
  Second modality is defined as laser photocoagulation, episcleral buckling, vitrectomy, and anti-VEGF therapy with different type of drug from the first treatment.

OTHER OUTCOMES:
VEGF levels in the systemic circulation | Before the first treatment (Day 0), Day 1, Week 1 and Week 24
  Blood samples for the determination of systemic VEGF levels were collected at the following time points: before the first treatment, at Day 1, at Week 1 and Week 24.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Department of Ophthalmology, the Second Affiliated Hospital of Xi'an Medical University, Xi'an, Shaanxi
  - Department of Ophthalmology, Xijing Hospital, Air Force Military Medical University, Xi'an, Shaanxi
  - Department of Ophthalmology, Xianyang Rainbow Hospital, Xianyang, Shaanxi